CLINICAL TRIAL: NCT06272734
Title: Reprieve System for the Treatment of Subjects With Acute Decompensated Heart Failure Pilot Study
Brief Title: Reprieve System Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reprieve Cardiovascular, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCV-0007
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Reprieve System (Experimental): Subjects will receive personalized and optimized diuretic and saline infusion using the study device during the course of the treatment.
  Interventions: Device: Reprieve System

INTERVENTIONS:
Device: Reprieve System — The study is broken into stages:
  1. In Stage one, Subjects enrolled in the study received Reprieve System (RS) therapy, a hospital bedside fluid management system designed to provide personalized and automated infusion of the IV diuretic furosemide and physiological saline in response to the patient's real-time urine output to safely and rapidly decongest patients suffering from Acute Decompensated Heart Failure. (complete, N=10)
  2. In future Stages, Subjects enrolled in the study will receive RS therapy and will be given varying levels of water consumption to challenge the algorithm. Future Stages will also assess new RS hardware and software features.

SUMMARY:
The objective of the study is to evaluate the use of the Reprieve System to decongest subjects with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a diagnosis of heart failure as defined by the presence of at least 1 symptom (dyspnea, orthopnea, or edema/swelling) AND 1 sign (peripheral edema, ascites, jugular venous distension, pulmonary vascular congestion on chest radiography)
2. ≥10 lb. (4.5 kg) above dry weight either by historical weights or as estimated by health care provider.
3. Patients ≥ 18 years of age able to provide informed consent and comply with study procedures.

Exclusion Criteria:

1. Inability to place Foley catheter or IV catheter or other urologic issues that would predispose the patient to a high rate of urogenital trauma or infection with catheter placement.
2. Hemodynamic instability as defined by any of the following: systolic blood pressure <90 mmHg, use of vasopressors, use of IV inotropes to treat hypotension (systolic blood pressure <90 mm Hg) or suspected/confirmed low cardiac output/shock, mechanical circulatory support, uncontrolled arrhythmias, active severe bleeding, or confirmed or suspected cardiogenic shock. Note: In the absence of the above conditions, use of inotropes to augment diuresis is permitted.
3. Dyspnea due primarily to non-cardiac causes (e.g., severe chronic obstructive pulmonary disease or pneumonia).
4. Acute infection with evidence of systemic involvement (e.g., clinically suspected infection with fever or elevated serum white blood cell count).
5. Estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2 calculated using the MDRD equation or current use of renal replacement therapy (RRT).
6. Significant left ventricular outflow obstruction, uncorrected complex congenital heart disease, known severe stenotic valvular disease, infiltrative or constrictive cardiomyopathy, acute myocarditis, type 1 acute myocardial infarction requiring treatment (within previous week), or any other pathology that, in the opinion of the investigator, would make aggressive diuresis poorly tolerated.
7. Inability to follow instructions or comply with follow-up procedures.
8. Other concomitant disease or condition that investigator deems unsuitable for the study, including drug or alcohol abuse or psychiatric, behavioral, or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the protocol instructions or follow-up procedures.
9. Severe baseline electrolyte abnormalities (e.g., serum potassium <3.0 mEq/L or magnesium <1.3 mEq/L). Note: These are based on baseline/screening labs. Subjects whose electrolyte levels are repleted cannot be reassessed for inclusion in the trial.
10. Serum sodium <135 mmol/L or history of severe hyponatremia
11. Poorly controlled diabetes
12. Enrollment in another interventional trial during the index hospitalization
13. Life expectancy less than 3 months
14. Women who are pregnant or intend to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Device Success | Over the 72-hours maximum duration of therapy.
  Defined as the device's ability to perform its intended function as specified in the study protocol without any device-related adverse events or malfunctions as determined by the treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Tamaz Shaburishvili, MD, Principal Investigator — Tbilisi Heart and Vascular Clinic
Locations (1):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No